CLINICAL TRIAL: NCT03841266
Title: Postoperative Recurrence Risk Evaluation of Hormone Receptor Positive, Her-2 Negative Breast Cancer by Using Different 21-gene Detection Kits (REBCK)
Brief Title: Recurrence Risk Evaluation by 21-gene Detection
Status: Completed | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, LiNanlin,Ph.D, Chief Physician,Clinical Professor, Professor, Thyroid breast and vascular surgery, Principal Investigator, Xijing Hospital
Other Study IDs: KY2019
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Relationship and Consistency Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: recurrence risk evaluation — Recurrence score were obtained by 21-gene detection kits from different biological companies. The expression of ER, PR, and Her-2 were also detected by IHC.

SUMMARY:
Breast cancer patients with early breast cancer were enrolled according to the inclusion criteria. Baseline characteristics were recorded from medical record system. Recurrence score were obtained by 21-gene detection kits from different biological companies. Relationship between recurrence score and the prognosis was explored. Meanwhile, the investigators analyzed the consistency of the results obtained from various 21-gene test kits and immunohistochemistry detection.

ELIGIBILITY:
Inclusion Criteria:

1. breast cancer in stage I-III, tumor size>0.5cm
2. lymph nodes negative
3. hormone receptor positive （ER+/PR+,ER+/PR-,ER-/PR+）
4. HER2 negative（IHC 0 or +， FISH negative）
5. receive endocrine therapy only
6. enough FFPE samples within 10 years（3~6 10μm ）
7. patients with integrated medical records

Exclusion Criteria:

1. Tumor cells <5%
2. Isolated RNA<500ng

Ages: 18 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients with early breast cancer were enrolled according to the inclusion criteria. Baseline characteristics were recorded from medical record system. Recurrence score were obtained by 21-gene detection kits from different biological companies. Relationship between recurrence score and the prognosis was explored. Meanwhile, we analyzed the consistency of the results obtained from various 21-gene test kits and immunohistochemistry detection.
Sampling Method: Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-01-20 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
correlation analysis | Janyary 1, 2019-December 31, 2019
  x2 value and P value of chi-square test

SECONDARY OUTCOMES:
consistency analysis | Janyary 1, 2019-December 31, 2019
  kappa value, P value of consistency analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing hoapital, Xi'an, China